CLINICAL TRIAL: NCT05863650
Title: The Effect of Digital-Based Simulation Education on Self-Efficacy and Clinical Reasoning Skills in Physiotherapy and Rehabilitation Students
Brief Title: The Effect of Digital-Based Simulation on Physiotherapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 22112022-108
Record Dates: First submitted 2023-04-27; First posted 2023-05-18 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-12

CONDITIONS: Self-efficacy; Clinical Reasoning
Keywords: Digital based simulation; Face to face education; Physiotherapy and rehabilitation students

STUDY DESIGN:
Intervention Model Description: Stepped wedge design
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Education (Experimental): 60 volunteer students participating in the study will start face-to-face training after preliminary evaluations are made. Afterwards, a randomized group of 10 people will be included in the simulation training every week. In the face-to-face education group, a case analysis will be applied by the students themselves together with the educators in the classroom environment. In the simulation group, one case analysis will be made every week on the website designed under the supervision of researchers.
  Interventions: Device: Digital based simulation
- Face to Face Education (Active Comparator): 60 volunteer students participating in the study will start face-to-face training after preliminary evaluations are made. Afterwards, a randomized group of 10 people will be included in the simulation training every week. In the face-to-face education group, a case analysis will be applied by the students themselves together with the educators in the classroom environment. In the simulation group, one case analysis will be made every week on the website designed under the supervision of researchers.
  Interventions: Other: Face to face education

INTERVENTIONS:
Device: Digital based simulation — Algorithms will be created for various musculoskeletal diseases and these algorithms will be controlled by taking the opinions of physiotherapists and physicians who are experts in their fields. After the algorithms are created, a website with patient scenarios containing these algorithms will be established with the support of a software company. In addition to the website, a database will be created and the applications made on the site will be recorded. In this way, the data of users using the website will be collected.
  Arms: Hybrid Education
Other: Face to face education — In the face-to-face education group, one case analyzes will be applied by the students together with the educators themselves in the classroom environment, with the educational content prepared in parallel with the patient scenarios in the simulation-based education group.
  Arms: Face to Face Education

SUMMARY:
In physiotherapy and rehabilitation education, basic medical courses, clinical information, rehabilitation approaches, special teachings of the profession, clinical problem solving and analysis in their fields are taught during university education.

Musculoskeletal problems will be selected for the patient scenarios to be used in the simulation and algorithms will be arranged for the simulation. After the algorithms are created, a website with patient scenarios containing these algorithms will be established with the support of a software company. In addition to the website, a database will be created and the applications made on the site will be recorded.

In our study, stepped wedge design will be used. 100 volunteer students participating in the study will start face-to-face training after preliminary evaluations are made. Afterwards, every two weeks, a randomized group of 20 people will be included in the hybrid training, which includes both face-to-face and simulation training. In the face-to-face education group, the educational content prepared in parallel with the patient scenarios in the hybrid education group will be applied in the classroom environment by the students together with the educators themselves. In the hybrid training group, one case analysis will be done every week on the website designed under the supervision of researchers, and one case analysis will be done through face-to-face training.

The self-efficacy and clinical reasoning levels of the students included in the study will be evaluated with the Physiotherapist Self-Efficacy Questionnaire and the Clinical Reasoning Assessment Tool. The same evaluations will be repeated after the students in both groups have completed their 10-week education. Afterwards, students' satisfaction levels and suggestions from the simulation will be evaluated with qualitative questions, and opinions and suggestions about simulation will be collected by creating themes.

DETAILED DESCRIPTION:
Clinical reasoning is one of the most fundamental skills in health professions education and is essential for engaging in clinical practice. In many studies, it is stated that the learning of the clinical reasoning process in undergraduate students should be included in the curricula and learning objectives.

Self-efficacy is a concept that is effective in shaping one's behavior. Academic self-efficacy is the individual's belief in himself about how successful he will be in the face of the academic tasks he will face throughout his academic life and at what level he can fulfill these tasks.

In recent years, digital learning designs have been increasingly used in teaching practices in higher education. Various designs offer opportunities to improve self-regulation abilities, facilitate active learning, and make the learning process more transparent. It covers a variety of technologies such as digital learning designs, virtual reality, podcasts, apps, educational games, 360° video and animations. These technologies can be applied directly in learning activities or combined with other planned learning activities.

In studies, digital learning designs in physiotherapy education have been criticized because they are not based on a theoretical learning perspective. A systematic review on the role of computer-assisted learning in physiotherapy education concluded that it has been substantially less researched compared to other health professions education.

ELIGIBILITY:
Inclusion Criteria:

* Being an undergraduate student at Marmara University Faculty of Health Sciences Physiotherapy and Rehabilitation Department
* Having agreed to participate in the study
* Being in the 6th semester of their studies

Exclusion Criteria:

* Refusing to participate in the study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-11 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Self-efficacy will be measured using a Turkish version of Physiotherapist Self-Efficacy Questionnaire-musculoskeletal area. | 6 weeks
  The questionnaire consists of 13 items. The participants will asked to indicate their confidence to perform the described task (1 = very little confidence; 5 = a lot of confidence). Higher scores are related more confidence self-efficacy.
  Outcomes will be evaluated before and after the intervention.
The 'Clinical Reasoning Assesment Tool (CRAT)' will be used in clinical reasoning assessment. | 6 weeks
  The CRAT, a rubric scale, is scored by the evaluator marking on the Visual Analog Scale. CRAT aims to assess students' readiness to enter the clinical setting and facilitate student self-monitoring. The tool aims to actively participate in the student's development by identifying strong or weak areas in three areas (content knowledge - procedural knowledge and psychomotor skill - conceptual reasoning).
  Outcomes will be evaluated before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montpetit-Tourangeau K, Dyer JO, Hudon A, Windsor M, Charlin B, Mamede S, van Gog T. Fostering clinical reasoning in physiotherapy: comparing the effects of concept map study and concept map completion after example study in novice and advanced learners. BMC Med Educ. 2017 Dec 1;17(1):238. doi: 10.1186/s12909-017-1076-z. PMID 29191189
- [Background] Zimmerman BJ. Self-Efficacy: An Essential Motive to Learn. Contemp Educ Psychol. 2000 Jan;25(1):82-91. doi: 10.1006/ceps.1999.1016. PMID 10620383
- [Background] Veneri D. The role and effectiveness of computer-assisted learning in physical therapy education: a systematic review. Physiother Theory Pract. 2011 May;27(4):287-98. doi: 10.3109/09593985.2010.493192. Epub 2010 Aug 8. PMID 20690881
- [Background] Odegaard NB, Myrhaug HT, Dahl-Michelsen T, Roe Y. Digital learning designs in physiotherapy education: a systematic review and meta-analysis. BMC Med Educ. 2021 Jan 13;21(1):48. doi: 10.1186/s12909-020-02483-w. PMID 33441140
- [Background] Blackstock FC, Watson KM, Morris NR, Jones A, Wright A, McMeeken JM, Rivett DA, O'Connor V, Peterson RF, Haines TP, Watson G, Jull GA. Simulation can contribute a part of cardiorespiratory physiotherapy clinical education: two randomized trials. Simul Healthc. 2013 Feb;8(1):32-42. doi: 10.1097/SIH.0b013e318273101a. PMID 23250189
- [Background] Sandoval-Cuellar C, Alfonso-Mora ML, Castellanos-Garrido AL, Del Pilar Villarraga-Nieto A, Goyeneche-Ortegon RL, Acosta-Otalora ML, Del Pilar Castellanos-Vega R, Cobo-Mejia EA. Simulation in physiotherapy students for clinical decisions during interaction with people with low back pain: randomised controlled trial. BMC Med Educ. 2021 Jul 9;21(1):375. doi: 10.1186/s12909-021-02812-7. PMID 34243767
- [Background] Zhong BL, Luo W, Li HM, Zhang QQ, Liu XG, Li WT, Li Y. Knowledge, attitudes, and practices towards COVID-19 among Chinese residents during the rapid rise period of the COVID-19 outbreak: a quick online cross-sectional survey. Int J Biol Sci. 2020 Mar 15;16(10):1745-1752. doi: 10.7150/ijbs.45221. eCollection 2020. PMID 32226294
- [Background] van Lankveld W, Jones A, Brunnekreef JJ, Seeger JPH, Bart Staal J. Assessing physical therapist students' self-efficacy: measurement properties of the Physiotherapist Self-Efficacy (PSE) questionnaire. BMC Med Educ. 2017 Dec 12;17(1):250. doi: 10.1186/s12909-017-1094-x. PMID 29233154
- [Background] Phillips AC, Mackintosh SF, Bell A, Johnston KN. Developing physiotherapy student safety skills in readiness for clinical placement using standardised patients compared with peer-role play: a pilot non-randomised controlled trial. BMC Med Educ. 2017 Aug 10;17(1):133. doi: 10.1186/s12909-017-0973-5. PMID 28797260
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Result] Holdar U, Wallin L, Heiwe S. Why do we do as we do? Factors influencing clinical reasoning and decision-making among physiotherapists in an acute setting. Physiother Res Int. 2013 Dec;18(4):220-9. doi: 10.1002/pri.1551. Epub 2013 May 2. PMID 23637022
- [Result] Torres G, Villagran I, Fuentes J, Araya JP, Jouannet C, Fuentes-Lopez E. Interactive virtual scenarios as a technological resource to improve musculoskeletal clinical reasoning skills of undergraduate physiotherapy students. Physiother Theory Pract. 2022 Aug;38(8):1016-1026. doi: 10.1080/09593985.2020.1809043. Epub 2020 Aug 19. PMID 32814476
- [Result] Hough J, Levan D, Steele M, Kelly K, Dalton M. Simulation-based education improves student self-efficacy in physiotherapy assessment and management of paediatric patients. BMC Med Educ. 2019 Dec 16;19(1):463. doi: 10.1186/s12909-019-1894-2. PMID 31842864
- [Result] Koivisto JM, Haavisto E, Niemi H, Haho P, Nylund S, Multisilta J. Design principles for simulation games for learning clinical reasoning: A design-based research approach. Nurse Educ Today. 2018 Jan;60:114-120. doi: 10.1016/j.nedt.2017.10.002. Epub 2017 Oct 24. PMID 29096383
- [Result] Halabchi F, Hassabi M. Acute ankle sprain in athletes: Clinical aspects and algorithmic approach. World J Orthop. 2020 Dec 18;11(12):534-558. doi: 10.5312/wjo.v11.i12.534. eCollection 2020 Dec 18. PMID 33362991